CLINICAL TRIAL: NCT00305175
Title: Long Term Effects of Hydroxyurea Therapy in Children With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: HUSTLE
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxyurea; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Prior Hydroxyurea: Patients who have received hydroxyurea therapy before entering the study.
- Patients Without Prior Hydroxyurea: Patients who have not received hydroxyurea before study entry.

SUMMARY:
The primary objectives of this prospective, observational study are (1) to describe the long-term cellular, molecular, and clinical effects of hydroxyurea therapy in sickle cell disease, and (2) to perform hydroxyurea pharmacokinetics studies.

This study will follow sickle cell patients being treated with hydroxyurea for a long period of time to evaluate the long-term cellular and molecular effects of the drug on the patients' body. This study will consist of two patient groups. One group will be made up of patients who have received hydroxyurea therapy before entering the study. The second group will be made up of patients who have not received hydroxyurea before study entry.

DETAILED DESCRIPTION:
Many years of study have documented the severe effects of sickle cell disease. Some of these effects include hemolysis (the break down of red blood cells), blockages in the blood vessels, and damage to the organs systems of the body. Hydroxyurea, which is given by mouth, is used to effectively prevent blockages in the blood vessels of patients with sickle cell disease. The hydroxyurea dosage varies and the responses of the body to this drug are not well understood.

This study will follow sickle cell patients being treated with hydroxyurea for a long period of time to evaluate the long-term cellular and molecular effects of the drug on the patients' body. This study will consist of two patient groups. One group will be made up of patients who have received hydroxyurea therapy before entering the study (Old Cohort). The second group will be made up of patients who have not received hydroxyurea before study entry (New Cohort).

This is not a therapeutic drug trial. Subjects for this study will receive hydroxyurea therapy for accepted clinical indications, and will be treated per best clinical management using treatment algorithms established at St. Jude Children's Research Hospital and other pediatric sickle cell programs across the United States. Hydroxyurea therapy data (such as dosing and duration of therapy) will not be dictated by this study, but will be collected to correlate with long-term outcomes. Hydroxyurea dose escalation to a stable MTD will occur according to published guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients from birth up to age 30 years
* Diagnosis of sickle cell disease
* Patients who are receiving hydroxyurea therapy or plan to begin hydroxyurea therapy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study participants will be patients with sickle cell disease who receive medical care from the Department of Hematology staff of St. Jude Children's Research Hospital. All patients on hydroxyurea therapy or patients who are initiating hydroxyurea therapy will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2006-03-03 (Actual); Primary Completion 2015-04-23 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
DNA damage from hydroxyurea therapy-variable-diversity-joining (VDJ) recombination events defined as the number of events per microgram of genomic DNA; | Every 3 years
DNA damage from hydroxyurea therapy-percentage of HJB in immature (CD71+) erythrocytes | Every 3 years

SECONDARY OUTCOMES:
Brain function as measured by MRI/MRA and TCD | Every 3 years
  optional test
Splenic function as measured by Spleen Scan | Every 3 years
  optional test
Kidney function as measured by BUN/creatinine and Urinalysis, glomerular filtration rate (GFR) | Every 3 years
  optional test
Lung function as measured by forced vital capacity (FVC) (%), forced vital volume in 1 second (FVC1) (%), and tricuspid regurgitation (TR) jet on Echocardiogram (ECHO) | Every 3 years
  collected if performed for clinical purposes
Growth as measured by height and weight | Every visit

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Estepp, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Power-Hays A, McElhinney KE, Williams TN, Mochamah G, Olupot-Olupot P, Paasi G, Reid ME, Rankine-Mullings AE, Opoka RO, John CC, McGann PT, Quinn CT, Punt NC, Smart LR, Stuber SE, Latham TS, Vinks AA, Ware RE. Hydroxyurea pharmacokinetics in children with sickle cell anemia across different global populations. Blood Adv. 2026 Jan 27;10(2):418-427. doi: 10.1182/bloodadvances.2025017254. PMID 41026975
- [Derived] Aygun B, Mortier NA, Smeltzer MP, Shulkin BL, Hankins JS, Ware RE. Hydroxyurea treatment decreases glomerular hyperfiltration in children with sickle cell anemia. Am J Hematol. 2013 Feb;88(2):116-9. doi: 10.1002/ajh.23365. Epub 2012 Dec 17. PMID 23255310
- [Derived] Flanagan JM, Steward S, Howard TA, Mortier NA, Kimble AC, Aygun B, Hankins JS, Neale GA, Ware RE. Hydroxycarbamide alters erythroid gene expression in children with sickle cell anaemia. Br J Haematol. 2012 Apr;157(2):240-8. doi: 10.1111/j.1365-2141.2012.09061.x. Epub 2012 Feb 24. PMID 22360576
- [Derived] Walker AL, Steward S, Howard TA, Mortier N, Smeltzer M, Wang YD, Ware RE. Epigenetic and molecular profiles of erythroid cells after hydroxyurea treatment in sickle cell anemia. Blood. 2011 Nov 17;118(20):5664-70. doi: 10.1182/blood-2011-07-368746. Epub 2011 Sep 14. PMID 21921042
- [Derived] Flanagan JM, Howard TA, Mortier N, Avlasevich SL, Smeltzer MP, Wu S, Dertinger SD, Ware RE. Assessment of genotoxicity associated with hydroxyurea therapy in children with sickle cell anemia. Mutat Res. 2010 Apr 30;698(1-2):38-42. doi: 10.1016/j.mrgentox.2010.03.001. Epub 2010 Mar 15. PMID 20230905
- See also: St. Jude Children's Research Hospital — http://stjude.org
- See also: Clinical Trials Open at St. Jude — http://stjude.org/protocols